CLINICAL TRIAL: NCT04307680
Title: Evaluation and Comparison of Short-term Efficacy Between Extracorporeal Magnetic Innervation and High-intensity Kegel Exercise Regimen
Brief Title: Evaluation and Comparison of Efficacy Between Extracorporeal Magnetic Innervation and High-intensity Kegel Exercise Regimen in Treatment of Stress Urinary Incontinence in Female
Acronym: KEMS-CRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Mislav Mikuš, Dr, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: UniZG
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel exercise (Active Comparator): Using high-intensity Kegel exercise regimen for 8 weeks (5 times a week; 3 times a day involved; 3 sets of 10-12 contractions)
  Interventions: Device: Peritron perineometer
- Magnetic stimulation (Active Comparator): Using 16 extracorporeal magnetic innervation treatments during 8 weeks (2 times a week).
  Interventions: Device: Peritron perineometer

INTERVENTIONS:
Device: Peritron perineometer — Perineometry will be used to assess quality of each observed treatment modality.

SUMMARY:
The aim of this prospective, randomized controlled study is to evaluate and compare efficacy between the most available conservative treatment (magnetic stimulation and Kegel exercise) for stress urinary incontinence in Croatia. We will assess quality-of-life, patient global improvement, and vaginal pressure measured with perineometer in three different time points: at the enrollment, after 8 weeks of treatment and 3 months after the both treatments are done.

ELIGIBILITY:
Inclusion Criteria:

* urodinamically confirmed stress urinary incontinence, at least one vaginal delivery in gynecological history.

Exclusion Criteria:

* urinary tract malignancies, vulvovaginitis, current uroinfection, previous pelvic surgeries, neurologic and psychiatric diseases, previous conservative treatment of stress urinary incontinence in less than 6 months, Stage III and IV of genital prolapse, latex allergy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-02 (Actual); Primary Completion 2021-01-02 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
Greater proportion of reduced ICIQ-SF score in magnetic stimulation arm group after 8 weeks of treatment | 8 weeks from the start of the treatment
  We assume that after 8 weeks of treatment, in magnetic stimulation arm of study, we will observe more treatment ''responders'' - with at least 4-point reduction in overall ICIQ-SF score

SECONDARY OUTCOMES:
Greater proportion of increased perineometry value in magnetic stimulation arm group | 8 weeks
  We assume that after 8 weeks of treatment, in magnetic stimulation arm of study, we will observe more treatment ''responders'' - at least more than 30% of increase in overall vaginal pressure, measured by a Peritron perineometer
Greater proportion of better patient global improvement in magnetic stimulation arm group | 3 months from treatment finish
  We assume that after 3 months of treatment finish, in magnetic stimulation arm of study, we will observe more women who are satisfied with the treatment, compared to Kegel exercise arm - using Patient Global Improvement Score (PGI-I)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Zagreb, Croatia, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From February 2021.